CLINICAL TRIAL: NCT05476146
Title: Re-routing of the Track in the Treatment of High Anal Fistula
Brief Title: Re-routing in Treatment High Anal Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Mohamed Abdelghany, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssutU
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rerouting of track of high anal fistula (Experimental)
  Interventions: Procedure: Rerouting of the track in high anal fitula

INTERVENTIONS:
Procedure: Rerouting of the track in high anal fitula — Treatment of high anal fistula by rerouting

SUMMARY:
The aim of this study is to evaluate the role of rereouting in treatment of high anal fistula and evaluate the success rate, the recurrence and incontinence and see if rerouting of the track is a good choice in treatment of high anal fistula?

DETAILED DESCRIPTION:
Anal fistula is a very common perianal condition associated with considerable morbidity and inconvenience to the patient. It is hollow tract lined with granulation tissue that connects an in-depth primary opening inside the anal canal to a superficial secondary opening in the perianal skin. It is mostly nonspecific infection of an anal gland in the intersphincteric space as the initiating pathology Different classifications have been put forward which categorize these Fistula into low or high simple or complex, or according to their anatomy into intersphincteric, trans-sphincteric, and supra-sphincteric or extra-sphincteric Surgical therapy is the main method used to treat anal fistula. The best treatment criterion is to eradicate the infected lesion, ensure sufficient drainage, and promote the closure of the fistula, while minimizing damage to the anal sphincter.

High anal fistulas require more complex treatment when compared to low anal fistula because of their complexity.

Rerouting is a transposition technique for the management of high anal and anorectal fistulae is described by Mann and Clifton in 1985. The method involves re-routing the extrasphincteric portion of the track into an intersphincteric position with immediate repair of the external sphincter. The newly posi-tioned intersphincteric fistula is then dealt with at a later date when the external sphincter is soundly healed .

The advantages of rerouting over other techniques in patients with high anal fistulae; patients had satisfactory results, decrease recurrence of fistulae or abscess formation. Healing is rapid, short hospital stay and continence to flatus and faeces preserved

ELIGIBILITY:
Inclusion Criteria:- patients with high anal fistula admitted at Asuit University Hospital at the period of study

Exclusion Criteria:- Any case with low anal fistula

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
evaluation the role of rerouting of the track in high anal fistula in treatemt | 6 months
  : collect result and see recurance and incontinence rate.